CLINICAL TRIAL: NCT02065024
Title: Food Matrix and Genetic Variability as Determinants of the Bioavailability and Biological Effects of a B-cryptoxanthin and Phytosterols-enriched Beverage; In Vitro and in Vivo Evaluation
Brief Title: Food Matrix and Genetic Variability as Determinants of Bioavailability and Biological Effects of Beta-cryptoxanthin and Phytosterols
Acronym: foodmagenpol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Fernando Granado Lorencio, dr Fernando Granado Lorencio, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: AGL2012-39503-C02-02
Record Dates: First submitted 2014-02-07; First posted 2014-02-17 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Hypercholesterolemia; Osteoporosis
Keywords: b-cryptoxanthin; plant sterols; serum Cholesterol; bone turnover markers
MeSH Terms: conditions — Hypercholesterolemia; Osteoporosis | interventions — Phytosterols

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- b-cryptoxanthin plus phytosterols (Active Comparator): Fruit and milk based beverage enriched with b-cryptoxanthin and phytosterols
  Interventions: Dietary Supplement: b-cryptoxanthin plus phytosterols
- control (Placebo Comparator): Fruit and milk based beverage not enriched
  Interventions: Dietary Supplement: b-cryptoxanthin plus phytosterols

INTERVENTIONS:
Dietary Supplement: b-cryptoxanthin plus phytosterols

SUMMARY:
Regular consumption of a beverage containing β-cryptoxanthin (b-Cx) and plant sterols (Ps) has been shown to exert a synergic effect in reducing cardiovascular risk and bone remodeling markers (formation and resorption). The present project aims to assess the influence of technological treatment and genetic variability on the bioavailability and the health effects of the added components (Ps, b-Cx), in particular to their potential role in prevalent disorders.In vitro and in vivo studies will be carried out to this effect. In vitro and in vivo studies (human intervention study) will be performed and cardiovascular, bone turnover and inflammation markers will be evaluated. Additionally, an in vitro colonic fermentation model and cell cultures will be used to explore anticarcinogenic effects and potential cytotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women; mild hypercholesterolemia

Exclusion Criteria:

* Use of cholesterol lowering drugs, hormonal therapy, vitamin and herbs supplements use

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
serum response of B-cryptoxanthin | 6 weeks of intervention
Serum response of phytosterols | 6 weeks

SECONDARY OUTCOMES:
Serum lipid profile | 6 weks of intervention
bone resorption markers | 6 weeks
interleukins | 6 weeks
Serum C-reactive protein | 6 weeks
Bone formation markers | 6 weeks
Sterols faecal levels | 6 weeks
Erythrocytes for eryptosis evaluation | 6 weeks

OTHER OUTCOMES:
Intestinal transporters polymorphisms, | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Puerta de Hierro-Majadahonda, Majadahonda (Madrid), Madrid, Spain

REFERENCES:
- [Derived] Cuevas-Tena M, Bermudez JD, Silvestre RLA, Alegria A, Lagarda MJ. Impact of colonic fermentation on sterols after the intake of a plant sterol-enriched beverage: A randomized, double-blind crossover trial. Clin Nutr. 2019 Aug;38(4):1549-1560. doi: 10.1016/j.clnu.2018.08.012. Epub 2018 Sep 7. PMID 30243503